CLINICAL TRIAL: NCT03515031
Title: Open Randomized Controlled Clinical Trial Comparing Oxygen Therapy by High Flow Nasal Cannulae and by Venturi Mask in the Treatment of Acute Respiratory Failure Due to Severe Pneumonia (Hi Flow Oxygen vs Venturi Mask In Pneumonia)
Brief Title: High Flow Nasal Cannulae vs Venturi Mask in Respiratory Failure Due to Pneumonia
Acronym: HiFlOViP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Roberto Cosentini, MD, Head of Emergency Room, Papa Giovanni XXIII Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PapaGiovanniH
Record Dates: First submitted 2018-04-11; First posted 2018-05-03 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Insufficiency; Pneumonia
Keywords: High Flow Nasal Cannula; Venturi mask
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia

STUDY DESIGN:
Intervention Model Description: open randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blind to the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula Oxygenation (Experimental): High Flow Nasal Cannula Oxygenation with a minimum flow ≥ 60L / min, and an FiO2 such as to maintain a SpO2 ≥ 92% for at least 48 hours until clinical stability
  Interventions: Device: High Flow Nasal Cannula Oxygenation
- Venturi Mask Oxygenation (Active Comparator): Venturi Mask Oxygenation, with an FiO2 such as to maintain an SpO2 ≥ 92% for at least 48 hours until clinical stability
  Interventions: Device: Venturi Mask Oxygenation

INTERVENTIONS:
Device: High Flow Nasal Cannula Oxygenation — Delivery of humidified and heated (37ºC) high flow oxygen
  Arms: High Flow Nasal Cannula Oxygenation
Device: Venturi Mask Oxygenation — delivery of high flow oxygen
  Arms: Venturi Mask Oxygenation

SUMMARY:
The primary objective of this study is to compare the efficacy of treatment with HFNC (group A) compared to administration of oxygen therapy by Venturi mask (group B, standard therapy) in terms of reaching of endotracheal intubation criteria during acute respiratory failure due to severe pneumonia.

Inclusion Criteria: Respiratory rate (RR) at rest ≥20 bpm or presence of respiratory distress (severe dyspnoea at rest or use of accessory respiratory muscles or abdominal paradox); PaO2 / FiO2 ≤250 during oxygenation with Venturi Oxygenation mask at FiO2 = 50% administered for at least 60 minutes; Diagnosis of pneumonia as the sole cause of acute respiratory failure. Randomization: 150 consecutive patients will be randomized either to High Flow Nasal Cannula Oxygenation (75 patients, HFNCO with flow ≥ 60 L/min and FiO2 to maintain SpO2 ≥ ) or Venturi Mask Oxygenation (control, 75 patients).

Patients from both groups will be treated with antibiotic therapy according to the IDSA/ATS 2007 guidelines for community-acquired pneumonia and the IDSA/ATS 2016 guidelines for hospital-acquired pneumonia.

Intubation Criteria:

MAJOR CRITERIA:

Cardiac or respiratory arrest Breathing pauses with loss of consciousness Severe hemodynamic instability Need for sedation

MINOR CRITERIA (maintained for ≥1h):

Reduction ≥30% of the value of the PaO2/FiO 2 compared to baseline Increased 20% if PaCO2 PaCO2 previous ≥40mmHg Worsening alertness as increased by one degree on the Kelly scale Persistence or onset of respiratory distress Vital parameters, Kelly scale and arterial blood gas analysis (BGA) will be performed on admission, and at 1, 24, at 48 hours, at the achievement of clinical stability, and whenever there is a clinical worsening.

Patients enrolled in HFNC arm will continue HFNC oxygenation until clinical stability, defined as:

Body temperature ≤ 37°C and ≥36°C for 24 consecutive hours Good ability in swallowing CRP and WBC normalization trend than the admission exams Hemodynamic stability Lack of respiratory distress SpO2 94-98% The primary outcome variable is the proportion of patients who reach the endotracheal intubation criteria - regardless of the actual intubation rate - within the first 48 hours of treatment. The primary analysis will be performed on the ITT population

DETAILED DESCRIPTION:
1.1 Basic information Pneumonia is still the most important infectious disease in terms of morbidity and mortality and is one of the most common causes of hospitalization for acute respiratory failure. The aim of this trial is to compare the use of High Flow Nasal Cannula (HFNC) oxygenation versus standard oxygen therapy in patients with hypoxemia due to pneumonia.

1.2 Rationale The oxygenation through HFNC allows the use of high concentrations of oxygen administered by a high gas flow, heated and humidified. This device allows both higher FiO2 and the presence of a positive end-expiratory pressure (PEEP) with a greater gas exchange.

2. Aims OF THE STUDY 2.1 Primary aim The primary aim of this study is to compare the efficacy of treatment with HFNC (group A) compared to administration of oxygen therapy by Venturi mask (group B, standard therapy) in terms of clinical failure during acute respiratory failure due to severe pneumonia 2.2 Secondary aims

The secondary aims are:

30-day mortality gas exchange improvement in-hospital length of stay adverse events as per prior

3. STUDY DESIGN 3.1 Design This is randomized, open, controlled, multicenter study 3.2 Number of patients The sample size is 150 patients. The enrolled subjects will be randomized in two Arms: Arm 1, intervention, 75 patients treated with HFNC, minimum flow ≥ 60L / min, FiO2 such as to maintain a SpO2 ≥ 92%, and Arm 2, reference technique, 75 patients treated with oxygen with Venturi mask, with FiO2 as to maintain a SpO 2 ≥ 92%.

3.3 Duration of the study The estimated time to complete the recruitment of cases is 24 months. Each subject will be followed from enrolment until discharge.

3.4 Evaluation 3.5.1 Primary endpoint The primary endpoint is the achievement of clinical failure defined as at least one major criteria Or

At least ≥2 of the minor criteria maintained for at least 1 consecutive hour:

MAJOR CRITERIA:

Cardiac or respiratory arrest Breathing pauses with loss of consciousness Severe hemodynamic instability Need for sedation

MINOR CRITERIA:

Reduction ≥30% of the value of the PaO 2 / FiO 2 compared to baseline Increased 20% if PaCO2 PaCO2 previous ≥40mmHg Worsening alertness as increased by one degree on the Kelly scale Persistence or onset of respiratory distress

3.5.2 Secondary endpoint

The secondary endpoint includes:

30 days mortality after admission. improvement of respiratory exchanges compared to baseline, rated at 1, 24 and 48 hours and at the achievement of clinical stability with arterial blood gas.

rate of adverse events length of hospital stay. 3.5.3 Follow-up At 30 days from admission, each subject will be assessed, possibly through telephone contact, to determine the status of life (secondary endpoint).

4. STUDIED POPULATION AND SELECTION CRITERIA 4.1 Examined population The studied population consists of individuals with pneumonia presenting to the Emergency Departments 4.2 Inclusion/exclusion criteria (see appropriate section)

5. SCREENING PROCEDURES, RANDOMISATION, MASKING 5.1 Randomization The statistician of the study will make randomization, preparing a list generated by the computer using a special program. The experimenter center will receive a group of envelopes progressively numbered, opaque, sealed in order to avoid any opening.

5.2 Masking This study is open, not being justified a possible double masking technique or sham procedures.

6. SCHEDULE AND STUDY PROCEDURES The study is divided into a baseline visit, followed by 1 visit at 1 hour, in the next 24 hours, followed by another visit during the 48-hour and the last when clinical stability is achieved The patient then will be followed until discharge and with a visit or a follow-up interview after 30 days of admission to determine the status of life.

6.1 Clinical evaluation

Clinical evaluations include:

collection of history (prior and concomitant diseases), and any concomitant therapies complete physical exam only at baseline respiratory symptoms at each evaluation vital signs during each evaluation dyspnea assessment at every clinical evaluation, using the Borg scale axillary body temperature (BT) every 8 hours Kelly scale assessment at each evaluation.

6.2 Laboratory evaluations Unless otherwise specified, the following tests will be performed on admission, 24 hours and then every 48 hours until discharge criteria are reached.

CBC: (5 mL in EDTA); Biochemistry: blood urea nitrogen, creatinine, serum sodium, potassium, glucose, ALT, AST, creatine phosphokinase (CPK), bilirubin, C-reactive protein, albumin (5 mL whole blood); lactates: performed at baseline and subsequent blood gas controls (3 mL of whole blood) pregnancy test on the urine sample (only at baseline) The arterial blood gas analysis (BGA) with the calculation of PaO2/FiO2 will be performed on admission, at 1, 24, at 48 hours, and at the achievement of clinical stability, and whenever there is a clinical worsening.

6.3 Instrumental exams Routine chest x-ray on admission, as well as whenever a clinical deterioration occurs.

6.4 Examinations plan 6.4.1 Baseline medical exam For each patient it will be made physical examination and lab evaluation as described previously Then it will proceed to randomization as indicated in § 5.2. 6.4.2 Treatment period The doctor in charge is free to perform all measurements, including BGA, as needed to assess the patient's condition. These will be in the clinic folder but they are not part of the data analyzed for the study, with the exception of blood gas analysis necessary to determine the minor intubation criteria (§ 3.5.1). Such measures will be noted for determination of primary endpoint, but they will not be used for the measurement of gas exchange trend (secondary endpoint).

For the analysis of secondary endpoint, after 24 hours, 48 hours and the achievement of clinical stability should be measured and recorded:

vital parameters (BP, HR, RR). The BT is measured every 8 hours with other vital parameters evaluation of dyspnea using both the Borg scale and the Kelly scale adverse events BGA during the treatment with lactate measurement (maintaining the HFNC and oxygen therapy with a mask as defined for randomization) and evaluation of P/F ratio, A-a difference of O2 and arterial O2 consumption.

24 hours after randomization there will be rated the severity score the SAPS-II scale and the SOFA score in case of sepsis.

Every 48 hours there will be performed blood samples (CBC, biochemistry, CRP) until the clinical stability is reached.

If intubation criteria are reached, the study must be regarded as concluded. For patients enrolled in HFNC arm, the ventilatory support therapy using HFNC must be continued until the clinical stability, considered as the fulfillment of the following clinical stability.

After attainment of all clinical stability, there will be an attempt to remove HFNC and to put the patient in Venturi mask, with the same FiO2 as the HFNC used before.

This step will be considered definitive when one hour after the attempt the SpO2 remains 94-98% and the absence of respiratory distress or FR <25 acts per minutes.

For patients in Venturi group, as soon as clinical stability is reached through the fulfillment of clinical stability criteria, the successive evaluation takes place at the time of discharge.

6.4.3 End-study medical examination The visit will take place at the end of the study at the time of discharge or when intubation criteria will be achieved.

Evaluation will include:

vital parameters (BP, HR, RR) respiratory symptoms using both the Borg and the Kelly scale SpO2 6.4.4 Observations to 30 days or in case of unplanned evaluation

After 30 days of enrolment the patient will be requested via telephone interview of the subject or of the reference family:

If the participant is alive any hospitalization

7. STUDIED TECHNIQUES The two techniques in this trial are widely known and used for oxygen therapy, although still lacks a comparative assessment of efficiency in the case examined in this study

8. ASSESSMENT OF SCIENTIFIC AIMS 8.1 See appropriate section on Outcome measures 9. STATISTICAL CONSIDERATIONS 9.1 Studied population The study population consists of adult and consenting subjects, from to the ER population diagnosed with pneumonia as the unique cause of acute respiratory and PaO2/FiO2 ≤ 250 during oxygen with Venturi mask with FiO2 50% administered for at least 60 minutes.

9.2 Study design The study follows the randomized, controlled design vs. standard open intervention. Randomization is defined by the main statistician. The center receives a set of disposable sealed envelopes, opaque, prepared by the main statistician in blocks in accordance with procedures stored by itself. Each subject enrolled will receive the treatment indicated inside the envelope with the lowest number available.

9.3 Outcome measures of the study See appropriate section on Outcome Measures

9.4 Study hypothesis The study aims to evaluate the null hypothesis according to the proportion of patients reaching the primary endpoint does not differ in its populations.

9.5 Sample size The aim of the study is the null hypothesis examination, which indicates that the groups in the two populations are the same.

With the proposed sample of 75 subjects in both the two groups (a total of 150 subjects), the study has a power of 80% to give statistically significant results. This calculation assumes that the proportion of subjects that reach the primary endpoint is approximately the 60% of the control group and that the treatment in question is able to reduce this proportion of 35%.

9.6 Patients enrolling and follow-up Overall, it is expected to enrol approximately 150 patients. The estimated duration of enrolment is about 12 months. Considering the period of follow up of the patients, the expected study duration is approximately 36 months.

9.7 Analysis plan 9.7.1 Primary variable analysis The primary variable is the proportion of patients who meet the criteria for endotracheal intubation - regardless of the actual intubation - during the treatment until the achievement of the clinical stability criteria. The primary analysis will be performed on the ITT population. The proportion of subjects qualified as a "failure" related to the achievement of the criteria for intubation will be analyzed by contingency tables (chi-square) accompanied by the confidence interval of the difference, by the relative risk estimates and by the NNT, if applicable. It may also be analyzed by multivariate logistic regression.

The proportion of subjects who achieved the outcome at a set time (secondary analysis), if relevant, will be tabulated by relative confidence intervals for the difference and estimated odds-ratios for daily intervals.

9.7.2 Secondary variables analysis The Secondary endpoints include both continuous and binary distribution variables. The 30-day mortality will be analyzed by contingency tables and using multivariate logistic regression, considering as membership population these three categories: HFNC, Venturi (if randomized to standard after treatment maintained until the end of observation) and Mixed (if randomized to standard treatment and subsequently transferred to HFNC before the observation term)

ELIGIBILITY:
Inclusion Criteria:

* male or female of any ethnic group
* age greater than or equal to 18 years;
* respiratory rate (RR) at rest ≥ 20 breaths/minute or presence of respiratory distress (severe - dyspnea at rest or use of accessory respiratory muscles or paradox abdominal movement) PaO 2/ FiO 2 ≤250 during oxygen therapy with Venturi mask with FiO 2 50% administered for at least 60 minutes;
* diagnosis of pneumonia as the unique cause of acute respiratory failure
* informed consent obtained from the patient or the closest relative in case of patient's inability to give it.

Exclusion Criteria:

* other diagnoses (instead of pneumonia) as a cause of acute respiratory failure
* unstable angina and acute myocardial infarction in place;
* Acute respiratory acidosis with pH <7.35 and PaCO 2 > 45 mmHg;
* systolic blood pressure <90 mmHg unresponsive to fluids or with amines
* severe arrhythmias;
* epileptic seizures;
* the degree of vigilance depending on the Kelly scale > 3 (see Appendix II)
* impaired swallowing, which increases the risk of pneumonia aspiration inability to protect airways
* craniofacial trauma or burns
* uncooperative patient
* presence of open wound (skull, chest, abdomen)
* respiratory arrest or need for intubation
* ongoing pregnancy or suspected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Failure | Participants will be followed for the duration of hospital stay, for a maximum of 30 days
  The primary endpoint is the achievement of clinical failure defined as:
  At least one of major criteria Or
  At least 2 or more of the minor criteria maintained for at least 1 consecutive hour:
  MAJOR CRITERIA:
  Cardiac or respiratory arrest Breathing pauses with loss of consciousness Severe hemodynamic instability (Heart Rate ≤ 50 bpm with loss of alertness or Systolic Blood Pressure ≤ 70 mmHg) Need for sedation
  MINOR CRITERIA (observed for ≥ 1 hour):
  Reduction ≥30% of the value of the PaO 2 / FiO 2 compared to baseline Increased 20% if PaCO2 PaCO2 previous ≥40mmHg Worsening alertness as increased by one degree on the Kelly scale (see Appendix II) Persistence or onset of respiratory distress ( severe dyspnea or use of accessories respiratory muscles or paradoxical abdominal motion)

SECONDARY OUTCOMES:
30-day mortality after admission | day 30
  mortality rate at 30 days after admission
improvement of respiratory exchanges compared to baseline | hospital admission (=day 1), day 2, until the achievement of clinical stability
  arterial blood gas evaluation of gas exchange and ventilation
adverse events | Hospital discharge; participants will be followed for the duration of hospital stay, an expected average of 1 week
  observation adverse events rate
hospital stay | Hospital discharge; participants will be followed for the duration of hospital stay, an expected average of 1 week
  length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: roberto cosentini, MD, Study Director — ASST Papa Giovanni XXIII, Bergamo, Italy
Locations (1):
- Vicky Rubini, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Liesching TN, Lei Y. Efficacy of High-Flow Nasal Cannula Therapy in Intensive Care Units. J Intensive Care Med. 2017 Jan 1:885066616689043. doi: 10.1177/0885066616689043. Online ahead of print. PMID 28110612
- [Background] Ischaki E, Pantazopoulos I, Zakynthinos S. Nasal high flow therapy: a novel treatment rather than a more expensive oxygen device. Eur Respir Rev. 2017 Aug 9;26(145):170028. doi: 10.1183/16000617.0028-2017. Print 2017 Sep 30. PMID 28794144
- [Background] Brambilla AM, Aliberti S, Prina E, Nicoli F, Del Forno M, Nava S, Ferrari G, Corradi F, Pelosi P, Bignamini A, Tarsia P, Cosentini R. Helmet CPAP vs. oxygen therapy in severe hypoxemic respiratory failure due to pneumonia. Intensive Care Med. 2014 Jul;40(7):942-9. doi: 10.1007/s00134-014-3325-5. Epub 2014 May 10. PMID 24817030
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577